CLINICAL TRIAL: NCT02359097
Title: High Resolution Steady State Blood Volume Maps in Glioblastoma Using MRI - A Multicenter Study
Brief Title: Steady State Blood Volume Maps Using Ferumoxytol Non-stoichiometric Magnetite MRI in Imaging Patients With Glioblastoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Edward Neuwelt, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB00009846; NCI-2015-00080 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SOL-13090-L; eIRB#9846; IRB00009846 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Ferrosoferric Oxide; gadoteridol; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Radiologists will be blinded to the type of cerebral blood volume (CBV) maps (steady state [SS] and dynamic susceptibility contrast [DSC]) and patient information.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (DSC/DCE-CBV, SS-CBV mapping) (Experimental): Patients receive 2 doses (2nd dose optional) of gadoteridol IV and undergo MRI including DSC or DCE-CBV mapping over approximately 45-60 minutes on day 1. Within 3 days, patients receive 3 doses of ferumoxytol non-stoichiometric magnetite IV and undergo MRI including DSC and SS-CBV mapping after each dose over approximately 90 minutes. Patients undergo MRI without contrast 24 hours after ferumoxytol non-stoichiometric magnetite over approximately 30 minutes. This 3 day series of imaging repeats at different stages of disease and may be performed up to 5 times: prior to surgery, prior to chemoradiation therapy, 4-6 weeks post-chemoradiation therapy, at time of progression on gadolinium MRI per RANO criteria, and again at time of progression (if the previous time of progression showed pseudoprogression).
  Interventions: Procedure: Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging; Drug: Ferumoxytol; Drug: Gadoteridol; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging — Undergo MRI including DSC or DCE-CBV mapping
  Other Names: DSC-MRI; Dynamic Susceptibility Contrast-Enhanced MRI; DYNAMIC SUSCEPTIBILITY-CONTRAST MRI
Drug: Ferumoxytol — Given IV
  Other Names: Feraheme; Ferumoxytol Non-Stoichiometric Magnetite
Drug: Gadoteridol — Given IV
  Other Names: Gadoteridolum; GD-HP-DO3A; HSDB 7549; ProHance; SQ 32692
Procedure: Magnetic Resonance Imaging — Undergo MRI including SS-CBV
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This clinical trial studies steady state blood volume maps using ferumoxytol non-stoichiometric magnetite magnetic resonance (MRI) in imaging patients with glioblastoma. MRI is a procedure in which radio waves and a powerful magnet linked to a computer are used to create detailed pictures of areas inside the body. Contrast agents, such as ferumoxytol non-stoichiometric magnetite, may enhance these pictures and increase visibility of tumor cells and the blood vessels in and around the tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Testing if steady state (SS)-cerebral blood volume (CBV) maps are superior to dynamic susceptibility contrast-(DSC)-CBV maps in visualizing of brain tumor blood volumes.

SECONDARY OBJECTIVES:

I. Development of the SS-CBV mapping for quantitative CBV estimation. II. Assessment of therapeutic response. III. Association with survival. IV. Correlation of relative cerebral blood volume (rCBV) with histology. V. Assessment of late ferumoxytol (ferumoxytol non-stoichiometric magnetite) enhancement at various stages of disease.

OUTLINE:

Patients receive 2 doses (2nd dose optional) of gadoteridol intravenously (IV) and undergo MRI including DSC or dynamic contrast enhanced imaging (DCE)-CBV mapping over approximately 45-60 minutes on day 1. Within 3 days, patients receive 3 doses of ferumoxytol non-stoichiometric magnetite IV and undergo MRI including DSC and SS-CBV mapping after each dose over approximately 90 minutes. Patients undergo MRI without contrast 24 hours after ferumoxytol non-stoichiometric magnetite over approximately 30 minutes. This 2-3 day series of imaging repeats at different stages of disease and may be performed up to 5 times: prior to surgery, prior to chemoradiation therapy, 4-6 weeks post-chemoradiation therapy, at time of progression on gadolinium MRI per Response Assessment in Neuro-Oncology (RANO) criteria, and again at time of progression (if the previous time of progression showed pseudoprogression).

After completion of study, patients are followed up at 2 and 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a known or presumed radiological diagnosis of glioblastoma (GBM); for presumed diagnosis of GBM, histological confirmation of GBM must be completed within 12 weeks of enrollment; (subjects will be removed from study and non-evaluable if no histologic diagnosis of GBM is confirmed)
* Subjects must be enrolled before starting chemoradiation, either pre -or post-surgery
* All subjects, or their legal guardians, must sign a written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization in accordance with institutional guidelines
* Sexually active women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; surgical intervention i.e. tubal ligation or vasectomy; post-menopausal > 6 months or abstinence) for at least two months after each cycle of the study; should a female become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

Exclusion Criteria:

* Subjects with clinically significant signs of uncal herniation, such as acute pupillary enlargement, rapidly developing motor changes (over hours), or rapidly decreasing level of consciousness, are not eligible
* Subjects with known allergic or hypersensitivity reactions to parenteral iron, parenteral dextran, parenteral iron-dextran, or parenteral iron-polysaccharide preparations; subjects with significant drug or other allergies or autoimmune diseases may be enrolled at the investigator's discretion
* Subjects who are pregnant or lactating or who suspect they might be pregnant
* Subjects who have a contraindication for 3 tesla (T) MRI: metal in their bodies (a cardiac pacemaker or other incompatible device), are severely agitated, or have an allergy to gadolinium containing contrast material
* Subjects with known iron overload (genetic hemochromatosis); in subjects with a family history of hemochromatosis, hemochromatosis must be ruled out prior to study entry with normal values of the following blood tests: transferrin saturation (TS) test and serum ferritin (SF) test; all associated costs will be paid by the study
* Subject who have received ferumoxytol within 3 weeks of study entry
* Subjects with three or more drug allergies from separate drug classes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-01-06 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Assessment of overlay accuracy with 3-dimensional (3D) anatomical T1w post contrast scans (MPRAGE) | Up to 6 weeks after last visit
  Will be analyzed and the mean score between the two readers will be used in the primary analyses. That is, to compare steady state-cerebral blood volume (SS-CBV) maps and dynamic susceptibility contrast (DSC)-CBV maps, a linear mixed effects model will be used to compare the mean of the visualization variables between SS and DSC overall and at each of time points (before chemoradiation, after chemoradiation, at progression and after second line treatment) while taking into account the correlation due to repeated measures, and the clustering within institutions. Model assumptions will be evaluated and alternative models will be explored as necessary.
Confidence in identifying the lesion corresponding areas on cerebral blood volume (CBV) maps | Up to 6 week after last visit
  Will be analyzed and the mean score between the two readers will be used in the primary analyses. That is, to compare steady state (SS)-CBV maps and dynamic susceptibility contrast (DSC)-CBV maps, a linear mixed effects model will be used to compare the mean of the visualization variables between SS and DSC overall and at each of time points (before chemoradiation, after chemoradiation, at progression and after second line treatment) while taking into account the correlation due to repeated measures, and the clustering within institutions. Model assumptions will be evaluated and alternative models will be explored as necessary.
Assessment of cerebral blood volume (CBV) in small (< 1 cm) enhancing lesions | Up to 6 weeks after the last visit
  Will be analyzed and the mean score between the two readers will be used in the primary analyses. That is, to compare steady state (SS)-CBV maps and dynamic susceptibility contrast (DSC)-CBV maps, a linear mixed effects model will be used to compare the mean of the visualization variables between SS and DSC overall and at each of time points (before chemoradiation, after chemoradiation, at progression and after second line treatment) while taking into account the correlation due to repeated measures, and the clustering within institutions. Model assumptions will be evaluated and alternative models will be explored as necessary.
Delineation of tumor from larger blood vessels | Up to 6 weeks after last visit
  Will be analyzed and the mean score between the two readers will be used in the primary analyses. That is, to compare steady state-cerebral blood volume (SS-CBV) maps and dynamic susceptibility contrast (DSC)-CBV maps, a linear mixed effects model will be used to compare the mean of the visualization variables between SS and DSC overall and at each of time points (before chemoradiation, after chemoradiation, at progression and after second line treatment) while taking into account the correlation due to repeated measures, and the clustering within institutions. Model assumptions will be evaluated and alternative models will be explored as necessary.

SECONDARY OUTCOMES:
Overall survival | Up to 6 weeks after last visit
  For the assessment of therapeutic response and association with survival, the cerebral blood volume (CBV) values will be correlated with survival using a Cox mixed effects regression model while adjusting patient demographical and clinical characteristics and the clustering within institutions. To determine at which stage of the disease the steady state CBV will best predict survival as well as the best cut off points, separate models will be fit for different disease stages and different cutoff points including 1.75, others and the Response Assessment in Neuro-Oncology (RANO) criteria.
Relative cerebral blood volume (rCBV) values | Up to 6 weeks after last visit
  A linear model will be used to assess correlation of rCBV with histology based on the availability of data.
Ferumoxytol enhancement | 24 hours after ferumoxytol administration
  A linear mixed effects regression model will first be used to examine the relationship between transverse relaxation rate and ferumoxytol doses while taking the correlation due to repeated measures into account. If the relationship between transverse relaxation rate and ferumoxytol doses does not show good linearity, alternative function forms will be tested, for example, polynomial or exponential.

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Neuwelt, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - OHSU Knight Cancer Institute, Portland, Oregon